CLINICAL TRIAL: NCT06889974
Title: Timing of Renal Replacement Therapy Initiation in Tumor Lysis Syndrome
Acronym: TENDERS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/104
Record Dates: First submitted 2025-02-25; First posted 2025-03-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Renal Replacement Therapy for Acute Kidney Injury in ICU
Keywords: tumoral lysis syndrome; acute kidney injury; renal replacement therapy, timing
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with early initiation of renal replacement therapy (RRT): Patients with early initiation of RRT, RRT within 24 hours of acute kidney injury (AKI) diagnosis.
- Patients with delayed initiation of RRT: Patients with delayed initiation of RRT, RRT initiated only after urgent clinical indications arise, such as severe hyperkalemia or metabolic acidosis.

SUMMARY:
The TENDERS study aims to evaluate the impact of the timing of renal replacement therapy (RRT) initiation on outcomes in patients with tumor lysis syndrome (TLS) and associated acute kidney injury (AKI). The study will compare early versus delayed RRT initiation, examining the effect on renal function at 30 days post-treatment.

DETAILED DESCRIPTION:
Tumor lysis syndrome (TLS) is a common and life-threatening complication in patients with hematologic malignancies, characterized by severe metabolic imbalances due to rapid tumor cell destruction. This syndrome frequently leads to acute kidney injury (AKI), requiring renal replacement therapy (RRT) in about 50% of cases. Despite its clinical significance, there is a lack of consensus on the optimal timing of RRT initiation in TLS-related AKI. Studies in other forms of AKI suggest no difference in outcomes between early and delayed RRT initiation, but these results are not directly applicable to TLS patients. This study seeks to fill this gap by analyzing the timing and outcomes of RRT initiation in TLS patients. The retrospective study will collect data from multiple intensive care units (ICUs) across France. Procedure: The study will retrospectively analyze patient data from 2013 to 2023, comparing early vs. delayed RRT initiation. Follow-up: Data on renal function, RRT usage, and mortality will be collected 30 days and one year after ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Hospitalized in the ICU between January 1, 2013, and December 31, 2023.
* Diagnosed with a hematologic malignancy or solid tumor requiring chemotherapy.
* Diagnosed with TLS based on the presence of two or more biochemical criteria (e.g., hyperkalemia, hyperphosphatemia, hyperuricemia, hypocalcemia) within 3 days before or 7 days after chemotherapy initiation.

Exclusion Criteria:

* Patient or family opposition to data collection for research purposes.
* Incomplete medical records that preclude data extraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective, multicenter cohort study conducted across several intensive care units (ICUs) in France. Data will be collected retrospectively from patient records and analyzed to assess the impact of early versus delayed RRT initiation on clinical outcomes in patients with TLS-induced AKI.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Renal dysfunction at ICU discharge | From baseline to up to 30 days .
  The primary outcome is renal dysfunction at ICU discharge, defined as a ≥25% increase in serum creatinine from baseline, assessed at the time of ICU discharge.

SECONDARY OUTCOMES:
Incidence of AKI | At baseline
  Incidence of AKI related to Tumor lysis syndrome (TLS), assessed at ICU admission.
Use of RRT for TLS-related AKI | From baseline to up to 30 days.
  Use of RRT for TLS-related AKI, assessed during ICU stay.
Renal recovery | At 90 days after baseline
  90-day renal recovery, assessed at 90 days post-admission.
Long-term renal function | 12 months after baseline
  Long-term renal function is assessed by creatinine at one year
Mortality at 30 days | 30 days after baseline
  Mortality rate at 30 days.
Mortality at 12 months | 12 months after baseline
  Mortality rate 12 months post ICU admission
Long-term renal function | 12 months after baseline
  Long-term renal function is assessed by glomerular filtration rate at one year

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU d'Angers, Angers
  - Hôpital Pellegrin, Bordeaux
  - Hôpital la cavale blanche, Brest
  - CHU Dupuytren 1, Limoges
  - Hôtel-Dieu, Nantes
  - CHR d'Orléans, Orléans
  - CH de Pau, Pau
  - Centre Urgences-Réanimations, Rennes
  - IUCT-O Hopital Purpan, Toulouse
  - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No